CLINICAL TRIAL: NCT06160726
Title: Evaluating the Validation of MRI-based Artificial Intelligence Software (NNS-SOT) for Onset Time Estimation in Lesion With Acute Ischemic Stroke : a Single-center, Single-arm, Single-blind (Evaluator), Retrospective Pivotal Trial
Brief Title: MRI-based Artificial Intelligence Software (NNS-SOT) for Onset Time Estimation in Lesion With Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Nunaps Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: NNS-SOT-01
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the efficacy of investigational device named Stroke Onset Time Artificial Intelligence(AI) (Model name:NNS-SOT). Using the investigational device, analyze the image and the onset time of occurrence of acute ischemic stroke lesion on the brain image (4.5 hours or more from the onset of symptoms) and evaluate the efficacy of correctly estimating the onset time.

DETAILED DESCRIPTION:
This clinical trial software medical device (Model name: NNS-SOT) is developed based on artificial intelligence algorithms.

Through clinical validation, it will be easier to determine whether the golden hour (4.5 hours) has elapsed at the time of cerebral infarction in the medical field. It can be used for estimation of the onset time of occurrence in acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Brain imaging in patients with acute ischemic stroke aged 20 years and older
* Brain imaging of ischemic stroke manifestation lesion confirmed by medical staff in brain MR image
* Brain imaging taken within 24 hours of ischemic stroke symptoms
* Brain imaging including Magnetic Resonance(MR) images (DWI and FLAIR)
* Patients with clearly recorded onset time of acute ischemic stroke symptoms

Exclusion Criteria:

* Brain imaging used in NNS-SOT development process
* Brain imaging with noise (Artifact)
* Brain images damaged in data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cerebral infarction disease Brain imaging data taken from 474 subjects who visited clinical trial institution (From 2017 to March 27, 2023)
Sampling Method: Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | October - November 2023
  Evaluation of sensitivity and specificity of clinical performance (estimation of 4.5 hours or more after cerebral infarction) performed with clinical trial medical device

SECONDARY OUTCOMES:
Area Under the Curve(AUC), which is the lower area of the Receiver Operating Characteristics(ROC) curve | October - November 2023
  Lower limit of 95% confidence interval is 80% or more

CONTACTS AND LOCATIONS:
Overall Officials: Bum Joon Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea